CLINICAL TRIAL: NCT06995209
Title: The Effect of Acute Pre-Workout Supplementation on Shooting Accuracy in Well-Trained Basketball Players
Brief Title: Study on How Pre-Workout Supplements Affect Shooting Accuracy in Trained Basketball Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Athanasios Douligeris, Principal Investigator, International Hellenic University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 38/24-23.04.2024
Record Dates: First submitted 2025-04-26; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Athletic Performance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Phase (Experimental): Participants receive placebo supplement
  Interventions: Dietary Supplement: Placebo
- Supplement Phase (Experimental): Participants receive the pre-workout supplement
  Interventions: Dietary Supplement: Pre-workout Supplement

INTERVENTIONS:
Dietary Supplement: Placebo — 20 g, ~74 Kcal, 97% flavored maltodextrin, similar in color, flavor, taste, and energy as PWS
  Arms: Placebo Phase
Dietary Supplement: Pre-workout Supplement — 20 g, ~73 Kcal, 200 mg caffeine, 3.3 g creatine monohydrate, 3.2 g β-alanine, 6 g citrulline malate, and 5 g branched chained amino acid (BCAA)
  Arms: Supplement Phase

SUMMARY:
Basketball is a popular team sport where athletes score points by successfully shooting the ball into the basket. Accuracy in shooting is crucial for players to score points effectively. Pre-workout supplements (PWS) have garnered interest from athletes and fitness enthusiasts due to the purported synergistic action of their ingredients which, when consumed before training, may help improve athletic performance. The acute effect of PWS or similar on the shooting accuracy of basketball athletes has not yet been investigated. Therefore, this study aimed to investigate the acute effect of a caffeine-based PWS (containing caffeine, creatine, β-alanine, citrulline malate, and BCAAs) on the stationary free throw, two-point, and three-point shooting accuracy in basketball players.

DETAILED DESCRIPTION:
According to a randomized, double-blind, crossover, research design, 12 active and well-trained male basketball players will be recruited. The sample will participate in three treatments: 1) no supplement; 2) PWS and 3) Placebo (PL). Three field-based basketball shooting tests (stationary free throw, stationary two-point, and three-point shots) will be performed to assess shooting accuracy . During the first visit, participants who met the inclusion criteria will visit our laboratory for health assessment/ screening. At the same time, after receiving a detailed verbal explanation and written instructions from our team's registered nutritionist, participants will be advised to follow the exact same diet one day before the subsequent trials, one week apart. During the second visit, all participants will arrive at the basketball court to execute the shooting tests in the following order: 1) the stationary free throw shooting test (S1P), 2) the stationary two-point shooting test (S2P), and 3) the stationary three-point shooting test (S3P). One week later, during the third visit, all players will return to the same basketball court. They will receive a single dose either PWS or PL 30 minutes prior to the evaluations. Participants and researchers will all blinded as to the type of supplement consumed. Following that, they will complete the same measurements in the same order as in the second visit. A week later all procedures will be repeated, and participants will receive the alternative supplement depending on randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants, 18+
2. Absence of drugs, abuse or medications, which are known to affect the shooting accuracy

Exclusion Criteria:

1. Restraining orthopedic/neuromuscular issues
2. Caffeine hypersensitivity
3. Consumption of more than three servings of coffee per day
4. Use of any supplement or steroids prior to the study
5. Use of creatine, β-alanine, citrulline malate or BCAA-protein supplementation at least six months before the initiation of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The stationary free-throw shooting test | At baseline (no supplement), 30 minutes after placebo ingestion, and 30 minutes after PWS ingestion
  Each player will complete three sets of ten free throws, with a three-minute rest between sets. Two other players will stood under the hoop and pass the ball to the shooter.
The stationary two-point shooting test | At baseline (no supplement), 30 minutes after placebo ingestion, and 30 minutes after PWS ingestion
  Each athlete should execute two stationary two-point shots from five different positions, a total of ten shots. Two other players will collect the ball and return it to the shooter. This procedure will be repeated three times, with three minutes rest between each round, resulting in a total of 30 shots. The average successful scoring percentage from the three trials will used for analysis.
The stationary three-point shooting test | At baseline (no supplement), 30 minutes after placebo ingestion, and 30 minutes after PWS ingestion
  Each athlete should execute two stationary three-point shots from five different positions placed 6.75 meters, a total of ten shots. Two other players will collect the ball and return it to the shooter. This procedure will be repeated three times, with three minutes rest between each round, resulting in a total of 30 shots. The average successful scoring percentage from the three trials will used for analysis.

SECONDARY OUTCOMES:
Height | Baseline (Pre-Intervention)
  Height to the nearest 0.1cm will be measured using a stadiometer (Leicester portable height measure, Tanita HR 001, Tokyo, Japan
Body Mass and Composition | Baseline (Pre-Intervention)
  Body mass will be measured using a calibrated digital scale to the nearest 0.1 kg, while body fat percentage, body fat mass, and fat-free mass will be analyzed via bioelectrical impedance analysis.
Blood Pressure | Baseline (Pre-Intervention)
  An upper-body blood pressure monitor will be used to measure resting blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Sousana K. Papadopoulou, Study Director — International Hellenic University
Locations (1):
- Sports Nutrition Laboratory, International Hellenic University, Greece, Thessaloniki, Greece